CLINICAL TRIAL: NCT02664883
Title: MDSC Clinical Assay for Cancer Detection and Monitoring in Renal Cell Carcinoma
Brief Title: Myeloid Derived Suppressor Cells Clinical Assay in Finding Kidney Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4K-14-4; NCI-2015-01559 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-15-00309; 4K-14-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subject; Metastatic Renal Cell Cancer; Recurrent Renal Cell Carcinoma; Stage I Renal Cell Cancer; Stage II Renal Cell Cancer; Stage III Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I (no cancer or hematuria): Patients with no evidence of cancer and no hematuria undergo collection of blood and urine samples at baseline and 2 months for analysis via the Flow Cytometry MDSC Clinical Assay
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Group II (localized RCC): Patients diagnosed with localized renal cell carcinoma undergo collection of blood and urine samples at baseline and after nephrectomy for analysis via the Flow Cytometry MDSC Clinical Assay. Patients also undergo CT or MRI within 30 days after nephrectomy.
  Interventions: Procedure: Computed Tomography; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging
- Group III (metastatic RCC): Patients diagnosed with metastatic renal cell carcinoma undergo collection of samples prior to baseline and then after 4 months of systemic treatment for analysis via the Flow Cytometry MDSC Clinical Assay. Patients also undergo CT or MRI after completion of 4 months of systemic treatment.
  Interventions: Procedure: Computed Tomography; Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Computed Tomography — Correlative studies
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
  Groups: Group II (localized RCC); Group III (metastatic RCC)
Other: Cytology Specimen Collection Procedure — Undergo collection of blood and urine samples
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Correlative studies
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
  Groups: Group II (localized RCC); Group III (metastatic RCC)

SUMMARY:
This pilot research trial studies the use of the Myeloid Derived Suppressor Cells Clinical Assay in finding and monitoring kidney cancer. Studying samples of blood and urine from patients with kidney cancer in the laboratory may aid doctors in the early detection of cancer, monitor tumor response to therapy, detect the presence of occult spreading of disease, and identify early return of disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate a novel clinical assay (Myeloid Derived Suppressor Cells [MDSC] Clinical Assay) to detect cancer associated immune cells in the peripheral blood of patients as a means to better detect and monitor malignant renal cell carcinoma in patients.

II. Determine mean MDSC level, intra-subject variability, and inter-subject variability for three groups of subjects with variable renal cell carcinoma disease status at baseline.

III. In patients with known localized renal cell carcinoma who undergo nephrectomy, determine the change in MDSC level from diagnosis to after nephrectomy.

IV. In patients with known metastatic renal cell carcinoma who undergo systemic treatment, determine the change in MDSC level from baseline to after treatment (4 months) and, secondarily, to compare these changes to the changes in tumor burden as evaluated by computed tomography (CT) scan or other imaging modality.

OUTLINE: Patients are assigned to 1 of 3 groups according to disease status.

GROUP I: Patients with no evidence of cancer and no hematuria undergo collection of blood and urine samples at baseline and 2 months for analysis via the Flow Cytometry MDSC Clinical Assay.

GROUP II: Patients diagnosed with localized renal cell carcinoma undergo collection of blood and urine samples at baseline and after nephrectomy for analysis via the Flow Cytometry MDSC Clinical Assay. Patients also undergo CT or magnetic resonance imaging (MRI) within 30 days after nephrectomy.

GROUP III: Patients diagnosed with metastatic renal cell carcinoma undergo collection of samples prior to baseline and then after 4 months of systemic treatment for analysis via the Flow Cytometry MDSC Clinical Assay. Patients also undergo CT or MRI after completion of 4 months of systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in this study must meet one of the 3 following criteria:

  * Group 1: Healthy individual with no history of cancer or hematuria
  * Group 2: Subject with a diagnosis of localized renal cell carcinoma (by imaging and eventual pathology) scheduled to undergo nephrectomy
  * Group 3: Subject with a diagnosis of metastatic renal cell cancer(by imaging and eventual pathology) who is scheduled to begin a new systemic therapy
* Any type of renal cell carcinoma (RCC); any prior therapy
* Performance status: 0-3
* Leukocytes >= 3,000/mcL (frequently used - numbers listed are examples, investigator should modify as needed)
* Absolute neutrophil count >= 1,500/mcL (frequently used - numbers listed are examples, investigator should modify as needed)
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* For normal subject arm: no evidence of cancer or hematuria
* For localized RCC arm: no evidence of metastatic disease, second cancer, prior chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* For metastatic RCC arm: no evidence of second cancer, prior chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* For all subjects: uncontrolled intercurrent illness including, but not limited to previous or current history of second malignancy unrelated to renal cell carcinoma; autoimmune disease or immune deficiency, chronic treatment with immunomodulatory therapies (e.g. glucocorticoids); significant trauma, surgery, or infection in the past two weeks or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with renal cell carcinoma and their accompanying partners who are seen at the Urologic Oncology and Medical Oncology Clinics of the Keck Medical Center of University Southern California (USC), Norris Cancer Center, and USC-Los Angeles County Hospital will be recruited for this trial.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
Change in MDSC level in patients with known metastatic renal cell carcinoma who undergo systemic treatment | Baseline to after 4 months of systemic treatment
  The change in MDSC level in patients with known metastatic renal cell carcinoma who undergo systemic treatment will be determined. These changes will be compared to the changes in tumor burden as evaluated by CT scan or other imaging modality.
Change in MDSC level in patients with localized renal cell carcinoma who undergo nephrectomy | Baseline to 30 days after nephrectomy
Mean MDSC level | Baseline
  The mean MDSC level, intra-subject variability, and inter-subject variability for three groups of subjects with variable renal cell carcinoma disease status will be determined at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States